CLINICAL TRIAL: NCT03468504
Title: Mirror Therapy and Treadmill Training for Patients With Chronic Stroke: A Pilot Randomised Controlled Trial
Brief Title: Mirror Therapy and Treadmill Training for Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Technology, Sligo (Other)
Responsible Party: Principal Investigator, Dr. John Bartlett, Head of Research, Institute of Technology, Sligo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITSligo
Record Dates: First submitted 2018-02-19; First posted 2018-03-16 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy; Exercise Test

STUDY DESIGN:
Intervention Model Description: Pilot Randomised Placebo Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Experimental Group saw mirror image of non-affected limb in mirror while walking on treadmill.
  Placebo Group saw no refection of the non-affected limb due to positioning of mirror while walking on treadmill.
  Outcome assessor was blinded to treatment allocation. They evaluated participants in separate lab and was asked not to discuss the treatment given to patients. Even if the patient mentioned the trials they would discuss the fact that they were using Mirrors and Treadmill.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy & Treadmill Training (Experimental): Mirror Therapy: Participants view a mirror reflection of their non-affected limb which is placed in their mid-sagittal plane for 30 mins per day, 3 days per week, for four weeks.
  Treadmill Training: Participants will walk on a treadmill at their comfortable walking speed for 30 mins per day, 3 days per week, for four weeks.
  Interventions: Device: Mirror Therapy; Device: Treadmill
- Placebo Mirror & Treadmill Training (Placebo Comparator): Placebo Mirror Therapy: Participants view a mirror which is placed forward/ahead of them in their mid-sagittal plane, and cannot see a reflection of any lower limb as their leg does not pass in front of the mirror for 30 mins per day, 3 days per week, for four weeks.
  Treadmill Training: Participants will walk on a treadmill at their comfortable walking speed for 30 mins per day, 3 days per week, for four weeks.
  Interventions: Device: Placebo Mirror Therapy; Device: Treadmill

INTERVENTIONS:
Device: Mirror Therapy — Participants view the reflective side of a simple mirror which is placed in their mid-sagittal plane to view a mirror reflection of their non-affected limb for 30 mins per day, 3 days per week, for four weeks.
  Other Names: Mirror Designed by IT Sligo.
  Arms: Mirror Therapy & Treadmill Training
Device: Placebo Mirror Therapy — Placebo Mirror Therapy: Participants view the reflective side of a simple mirror which is placed forward/ahead of them in their mid-sagittal plane, and thus cannot see a reflection of either lower limb as their leg does not pass in front of the mirror for 30 mins per day, 3 days per week, for four weeks.
  Treadmill Training: Participants will walk on a treadmill at their comfortable walking speed for 30 mins per day, 3 days per week, for four weeks.
  Other Names: Mirror Designed by IT Sligo.
  Arms: Placebo Mirror & Treadmill Training
Device: Treadmill — Participants will walk on a treadmill at their comfortable walking speed for 30 mins per day, 3 days per week, for four weeks.
  Other Names: Variable speed Treadmill.

SUMMARY:
This is a pilot randomised controlled trial investigating a combination of mirror therapy and treadmill training for the rehabilitation of lower limb impairment following a stroke. This study has been conducted as part of a PhD qualification at the Institute of Technology Sligo in Ireland with all therapy sessions taking place at the institute. The study was conducted in conjunction with Sligo University Hospital and it attained ethical approval through the relevant University Hospital Ethics Committee.

DETAILED DESCRIPTION:
The study necessitated patients with chronic stroke to walk on a treadmill while viewing a reflection of their non-affected limb in a mirror. There was also a placebo group and these patients walked on the treadmill and viewed a mirror in an altered position. Patients were referred through Hospital Health Professionals. Prior to trial commencement all participants were given comprehensive trial information and provided signed written informed consent. A total of 30 participants were recruited. Patients attended the study for 30 minutes per day, three days per week, for four weeks. Patients received outcome assessment prior to the beginning of the intervention, directly after it and at three month followup assessment. All assessments were carried out by a Chartered Physiotherapist specialising in stroke rehabilitation. Patients were assessed using established outcome measures for lower limb motor function, muscle tone, walking speed and endurance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke (greater than or equal to 6 months post stroke) with lower limb heimiparesis.
* Ambulatory with/without walking aid.
* Discharged from formal rehabilitation.
* A Mini Mental State Examination >/= 24.

Exclusion Criteria:

* Younger than 18 years
* Any additional illness that may prevent treadmill walking
* A Mini Mental State Examination < 24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Ten Metre Walk Test | 5 mins.
  Walking velocity measure. Lower times indicate an increased walking velocity.
Six Minute Walk Test | 10 mins
  Walking endurance measure. Larger distance indicates an improved walking endurance ability.

SECONDARY OUTCOMES:
Modified Ashworth Scale | 10 minutes
  Muscle tone measure. Range 0 (No increase in muscle tone) to 4 (Affected part(s) rigid in flexion or extension).
Fugl-Meyer Assessment-Lower extremity | 10 mins
  Motor function outcome. Range 0 (Unable to do any functional Task) to 34 (Fully Independent in Functional Lower Extremity Tasks).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Broderick, PhD, Principal Investigator — PhD researcher
Locations (1):
- Institute of Technology, Sligo, Sligo, Co Sligo, Ireland

IPD SHARING:
Plan to Share IPD: No
No IPD is shared with any other researchers.

DOCUMENTS (3):
  • Study Protocol (2014-12-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03468504/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03468504/SAP_001.pdf
  • Informed Consent Form (2014-12-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03468504/ICF_002.pdf